CLINICAL TRIAL: NCT05796674
Title: Post Market Clinical Follow-up (PMCF) Pilot Study for the Clareon UVA IOLs Using Retrospective Data Collection From the WaveTec AnalyzOR Database
Brief Title: Clareon IOL Retrospective Data Collection
Status: Completed | Type: Observational
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Other Study IDs: ILS241-R001
Record Dates: First submitted 2023-03-20; First posted 2023-04-03 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Aphakia; Astigmatism
MeSH Terms: conditions — Aphakia; Astigmatism | interventions — Drug Delivery Systems; Cataract Extraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Clareon UVA IOL: Eyes that underwent cataract surgery and received a Clareon UVA IOL with the use of the WaveTec Optiwave Refractive Analysis (ORA) System
  Interventions: Device: Clareon UVA IOL; Device: WaveTec Optiwave Refractive Analysis (ORA) System; Procedure: Cataract surgery

INTERVENTIONS:
Device: Clareon UVA IOL — Clareon UVA IOL placed in the capsular bag in the posterior chamber of the eye during cataract surgery to replace the natural crystalline lens. Models CC60WF and CCA0T0 are indicated for the visual correction of aphakia. Models CCW0T3, CCW0T4, CCW0T5, and CCW0T6 are indicated for the visual correction of aphakia and preexisting corneal astigmatism.
  Other Names: Models CC60WF, CCW0T3, CCW0T4, CCW0T5, CCW0T6, CCA0T0
Device: WaveTec Optiwave Refractive Analysis (ORA) System — Intra-operative system used during refractive cataract surgery to capture wavefront images of the patient's eye for the purpose of optimizing IOL implantation
Procedure: Cataract surgery — Cataract extraction by phacoemulsification, followed by implantation with a Clareon UVA IOL

SUMMARY:
The purpose of this study is to provide real world evidence (RWE) on the performance of the Clareon ultraviolet absorbing (UVA) intraocular lenses (IOLs) to support the overall body of evidence on the Clareon IOL family.

DETAILED DESCRIPTION:
In this retrospective postmarket study, the WaveTec AnalyzOR Database will be reviewed. All available data that meet the data selection criteria as of the data cutoff will be analyzed.

ELIGIBILITY:
Data Selection Criteria (eyes):

* Must have undergone cataract extraction by phacoemulsification with implantation of a Clareon UVA IOL (CC60WF, CCW0T3, CCW0T4, CCW0T5, CCW0T6, or CCA0T0) using the WaveTec ORA System.
* Must have a BCDVA in the WaveTec AnalyzOR Database from ≥ 10 days after surgery.
* Predicted residual refractive error spherical equivalent (SE) ≤ 0.75 D.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A description of the population from which the groups or cohorts will be selected (for example, primary care clinic, community sample, residents of a certain town).
  Information is entered into the WaveTec AnalyzOR Database by medical professionals post cataract surgery.
Sampling Method: Non-Probability Sample
Enrollment: 1090 (Actual)
Dates: Start 2023-08-18 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
Monocular Best Corrected Distance Visual Acuity (BCDVA) at Postoperative Visit | Month 1 postoperative
  The database will be reviewed for assessments of monocular (by-eye) best corrected distance visual acuity at the first postoperative visit. The first postoperative visit will be defined as the visit which occurred approximately 28 days or later from the operative visit during which time the IOL remained implanted in the eye and an eye exam was performed.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Lead, Surgical, Study Director — Alcon Research, LLC
Locations (1):
- Alcon Research, LLC, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No